CLINICAL TRIAL: NCT01007968
Title: A Phase I, Open-label, Multicenter Study to Evaluate the Pharmacokinetics and Safety of Oral Panobinostat in Patients With Advanced Solid Tumors and Various Degrees of Hepatic Function
Brief Title: Pharmacokinetics and Safety of Panobinostat in Patients With Advanced Solid Tumors and Various Degrees of Hepatic Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CLBH589X2101; 2009-012262-31 (EudraCT Number)
Record Dates: First submitted 2009-10-28; First posted 2009-11-05 (Estimated); Last update posted 2020-12-19 (Actual); Status verified 2016-08

CONDITIONS: Advanced Solid Tumors
Keywords: solid tumors; hepatic function; advanced; panobinostat
MeSH Terms: interventions — Panobinostat

ARMS (1):
- HDACi (Experimental)
  Interventions: Drug: LBH589

INTERVENTIONS:
Drug: LBH589

SUMMARY:
Panobinostat (LBH589) is a deacetylase inhibitor (DACi) which belongs to a structurally novel cinnamic hydroxamic acid class of compounds. It is one of the most potent class I/II pan-DAC inhibitor (pan-DACi) that has shown anti-tumor activity in pre-clinical models and patients with solid tumors and hematological malignancies.

To date, the pharmacokinetics (PK) of panobinostat has been characterized in patients with solid tumors and hematological malignancies participating in several phase I/II clinical studies. Panobinostat PK does not appear to be different in patients with solid tumors and hematological malignancies. However, the effect of organ dysfunction on PK of panobinostat is yet to be elucidated.

Kidney and liver are involved in the elimination and metabolism of panobinostat. The current study is designed to evaluate the impact of hepatic function status on panobinostat PK.

ELIGIBILITY:
Inclusion Criteria:

1. Patient has documented diagnosis of advanced solid tumor for which no standard systemic therapy exists
2. Patient has normal or abnormal hepatic organ function
3. Patient has provided written informed consent prior to any screening procedures

Exclusion Criteria:

1. Patient needing valproic acid for any medical condition during the study or within 5 days prior to the first panobinostat dose
2. Patient received prior treatment with DAC inhibitors including panobinostat
3. Patient requires treatment with warfarin that cannot be switched to another anticoagulant treatment prior to starting study drug
4. Patient has encephalopathy
5. Patient has ascites requiring intervention
6. Female patient who is pregnant or breast feeding or with childbearing potential and not willing to use a double method of contraception up to 3 months after the end of study treatment. Male patient who is not willing to use a barrier method of contraception up to 3 months after the end of study treatment.

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2010-03; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
To assess the effect of various degrees of impairment in hepatic function as measured by the National Cancer Institute-Cancer Therapy Evaluation Program (NCI-CTEP) criteria, on the pharmacokinetics of panobinostat. | first 7 days

SECONDARY OUTCOMES:
To assess the effect of various degrees of impairment in hepatic function on the safety of panobinostat | entire duration of study
To evaluate whether there is a relationship between panobinostat PK and safety parameters in patients with various degrees of hepatic organ function | first 7 days
To explore anti-tumor activity associated with panobinostat. | best overall response

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (6):
- University of Utah / Huntsman Cancer Institute, Salt Lake City, Utah, United States
- Novartis Investigative Site, Leiden, Netherlands
- Sweden (2):
  - Novartis Investigative Site, Lund
  - Novartis Investigative Site, Stockholm
- Novartis Investigative Site, Sankt Gallen, Switzerland
- Novartis Investigative Site, Edinburgh, United Kingdom

REFERENCES:
- [Derived] Slingerland M, Hess D, Clive S, Sharma S, Sandstrom P, Loman N, Porro MG, Mu S, Waldron E, Valera SZ, Gelderblom H. A phase I, open-label, multicenter study to evaluate the pharmacokinetics and safety of oral panobinostat in patients with advanced solid tumors and various degrees of hepatic function. Cancer Chemother Pharmacol. 2014 Nov;74(5):1089-98. doi: 10.1007/s00280-014-2594-6. Epub 2014 Sep 25. PMID 25253045
- See also: Results for CLBH589X2101 on the Novartis clinical trial website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=10384